CLINICAL TRIAL: NCT03004833
Title: Nivolumab and AVD in Early-stage Unfavorable Classical Hodgkin Lymphoma
Acronym: NIVAHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Paul Broeckelmann, Dr., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-2854
Record Dates: First submitted 2016-11-07; First posted 2016-12-29 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Nivolumab; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): 4 Cycles of Nivolumab plus AVD followed by IF-RT (30 Gy)
  Interventions: Drug: Nivolumab; Drug: Adriamycin; Drug: Vinblastine; Drug: Dacarbazine
- Arm B (Experimental): 4 Cycles of Nivolumab, followed by 2 cycles of Nivolumab plus AVD, followed by 2 Cycles of AVD followed by IF-RT (30 Gy)
  Interventions: Drug: Nivolumab; Drug: Adriamycin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Nivolumab — Infusion of Nivolumab
Drug: Adriamycin — Infusion of Adriamycin
Drug: Vinblastine — Infusion of Vinblastine
Drug: Dacarbazine — Infusion of Dacarbazine

SUMMARY:
The aim of the trial is to improve first-line treatment for early unfavorable cHL by introduction of the anti-PD-1 antibody Nivolumab with a truncated standard chemotherapy (AVD).

The primary objective is to show efficacy of the two experimental treatment strategies. Secondary objectives are to further evaluate efficacy, show safety and feasibility and perform correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven classical HL
* First diagnosis, no previous treatment
* Age: 18-60 years
* Stage I, IIA with risk factors a-d, IIB with RF c-d:

  1. large mediastinal mass
  2. extranodal lesions
  3. elevated ESR
  4. ≥ 3 nodal areas confirmed by central review.

Exclusion Criteria:

* Composite lymphoma or nodular lymphocyte- predominant Hodgkin lymphoma (NLPHL)
* History of other malignancy ≤ 5 years
* Prior chemotherapy or radiation therapy
* Concurrent disease precluding protocol treatment
* Pregnancy, lactation
* Non-compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Complete Remission Rate | 4 to 6 weeks after end of treatment

SECONDARY OUTCOMES:
Treatment related Morbidity | 1 year after end of treatment
Progression Free Survival | 1 and 3 years after end of treatment
Overall Survival | 1 and 3 years after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne, I. Dept. of Medicine
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brockelmann PJ, Buhnen I, Meissner J, Trautmann-Grill K, Herhaus P, Halbsguth TV, Schaub V, Kerkhoff A, Mathas S, Bormann M, Dickhut A, Kaul H, Fuchs M, Kobe C, Baues C, Borchmann P, Engert A, von Tresckow B. Nivolumab and Doxorubicin, Vinblastine, and Dacarbazine in Early-Stage Unfavorable Hodgkin Lymphoma: Final Analysis of the Randomized German Hodgkin Study Group Phase II NIVAHL Trial. J Clin Oncol. 2023 Feb 20;41(6):1193-1199. doi: 10.1200/JCO.22.02355. Epub 2022 Dec 12. PMID 36508302
- [Derived] Gerhard-Hartmann E, Goergen H, Brockelmann PJ, Mottok A, Steinmuller T, Grund J, Zamo A, Ben-Neriah S, Sasse S, Borchmann S, Fuchs M, Borchmann P, Reinke S, Engert A, Veldman J, Diepstra A, Klapper W, Rosenwald A. 9p24.1 alterations and programmed cell death 1 ligand 1 expression in early stage unfavourable classical Hodgkin lymphoma: an analysis from the German Hodgkin Study Group NIVAHL trial. Br J Haematol. 2022 Jan;196(1):116-126. doi: 10.1111/bjh.17793. Epub 2021 Sep 14. PMID 34520052
- [Derived] Brockelmann PJ, Goergen H, Keller U, Meissner J, Ordemann R, Halbsguth TV, Sasse S, Sokler M, Kerkhoff A, Mathas S, Huttmann A, Bormann M, Zimmermann A, Mettler J, Fuchs M, von Tresckow B, Baues C, Rosenwald A, Klapper W, Kobe C, Borchmann P, Engert A. Efficacy of Nivolumab and AVD in Early-Stage Unfavorable Classic Hodgkin Lymphoma: The Randomized Phase 2 German Hodgkin Study Group NIVAHL Trial. JAMA Oncol. 2020 Jun 1;6(6):872-880. doi: 10.1001/jamaoncol.2020.0750. PMID 32352505
- See also: Related Info — http://www.ghsg.org